CLINICAL TRIAL: NCT06914089
Title: Short and Long-term Outcomes of Biodegradable Coated Stent (Biomime Versus Ultimaster) Deployed in STEMI Patients Undergoing Primary Percutaneous Intervention
Brief Title: Thin Versus Thicker Strut Thickness Stents in Primary Percutaneous Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Ahmed Abdelnazeer, Short and long-term Outcomes of biodegradable coated stent (biomime versus ultimaster) deployed in STEMI patients undergoing primary percutaneous intervention, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Thin strut stents
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Primary Percutaneous Coronary Intervention
Keywords: primary percutaneous coronary intervention; ultrathin stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bio mime arm (Active Comparator): ultrathin stent arm
  Interventions: Device: The BioMime is an ultra-thin strut (65 µm) SES that uses a cobalt-chromium platform with a unique hybrid design of open cells in the mid segment and closed cells at the edges
- Ultimaster arm (Active Comparator): The Ultimaster® (Terumo CorporationTokyo, Japan) consists of the Kaname stent platform, abluminally coated with poly D,L-lactic acid-polycaprolactone (PDLLA-PCL) as a carrier of the immunosuppressant drug sirolimus (3.9 μg/mm stent length). The purpose of the gradient coating is to reduce potential cracking and delamination of the polymer. The drug release profile allows an initial stronger release immediately following stent implantation. Then the drug is released continuously until the polymer bioabsorption is completed within three to four months. For a stent size of 3.0×15 mm, the median maximum concentration (Cmax) was 36.8 pg/mL (range between 22.9 and 41.5 pg/mL), according to the previously published detailed information on the pharmacokinetic profile
  Interventions: Device: The BioMime is an ultra-thin strut (65 µm) SES that uses a cobalt-chromium platform with a unique hybrid design of open cells in the mid segment and closed cells at the edges

INTERVENTIONS:
Device: The BioMime is an ultra-thin strut (65 µm) SES that uses a cobalt-chromium platform with a unique hybrid design of open cells in the mid segment and closed cells at the edges — testing its safety and efficacy at long term follow up after primary percutaneous intervention

SUMMARY:
1. To evaluate clinical safety of the device in terms of Deaths, any stroke and Myocardial Infarction up to 1 year in both study groups to prove non inferiority of biomime stent
2. To evaluate presence of Target lesion and target vessel revascularization in in both study groups prove non inferiority of biomime stent
3. To evaluate target vessel non-target lesion revasularization in both study groups prove non inferiority of biomime stent

DETAILED DESCRIPTION:
• Drug-eluting stents (DES) represent a key advance in percutaneous coronary interventions (PCI) owing to their ability to inhibit neointimal proliferation, which lowers the need for repeat revascularisation However, older-generation DES have been shown to increase the risk of late restenosis and stent thrombosis. Efforts to reduce these risks include improvements in stent platforms, polymer carriers, and drug selection. Thinner struts reduce vessel wall injury, decrease inflammation and promote fast endothelialisation.The second-generation thin-strut DES have been shown to reduce the risk of restenosis, stent thrombosis and myocardial infarction (MI) or possibly death when compared with older-generation DES or bare metal stents. Moreover, the newer generation of biodegradable polymer stents has the potential to reduce the inflammatory reaction of the arterial wall and minimise the risk of late restenosis and thrombus formation More recently, ultra-thin (<70 μm) DES have been shown to improve outcomes further compared with second-generation DES.The BioMime™ (Meril Life Sciences Pvt. Ltd., Vapi, India) is an ultra-thin sirolimus-eluting coronary stent (SES) with an established preliminary safety and efficacy record in the previous meriT-1, meriT-2, meriT-3 and meriT-4 trials in treating single de novo and complex lesions.The BioMime is an ultra-thin strut (65 µm) SES that uses a cobalt-chromium platform with a unique hybrid design of open cells in the mid segment and closed cells at the edges which lead to Lesser Edge Dissections during expansion and Adequate Side Branch Access, coated with biocompatible and bioabsorbable polymers, PLLA (poly-L-lactic acid) and PLGA (poly-lactic-co-glycolic acid) for Faster Healing

ELIGIBILITY:
Inclusion criteria:

•All patients with ST-segment elevation myocardial infarction and diagnosed according to the last guidelines.

Exclusion Criteria:

* Left ventricular ejection fraction ≤30%.
* Killip class III or IV at presentation.
* Extreme vessel tortuosity or lesion angulation (˂45˚).
* Severe calcification proximal to or within the target lesion.
* Bifurcation lesions with side branch diameter >2 mm.
* Mechanical complication of STEMI.
* Severe comorbidity such as malignancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Target vessel failure | From enrollment and followed up for one year
  Target vessel failure (TVF): defined as cardiac death that cannot be clearly attributed to a vessel other than the target vessel, target vessel MI, and clinically driven target vessel revascularization
MACE | From enrollment and followed up for one year
  Major adverse cardiac events (MACE) as a composite of cardiac death, any MI and clinically driven target vessel revascularization (CD-TVR)
Late lumen Loss | From enrollment and followed up for one year
  Late lumen loss: the difference between the minimal luminal diameter (MLD) after stent implantation and after at least 9 months post procedure

SECONDARY OUTCOMES:
Device-oriented composite end points | From enrollment and followed up for one year
  Device-oriented composite end points (DOCE): Defined as Cardiovascular death, MI (not clearly attributable to a non-target vessel) and TLR (clinically driven)
Patient-oriented composite end points | From enrollment and followed up for one year
  Patient-oriented composite end points (POCE): Defined as all-cause mortality, any stroke, Any MI (includes non-target vessel territory) and Any revascularization
stent thrombosis | From enrollment and followed up for one year
  Definite stent thrombosis: The presence of a thrombus that originates in the stent or in the segment 5 mm proximal or distal to the stent or in a side branch originating from the stented segment and the presence of at least one of the following criteria:
  A) Acute onset of ischemic symptoms at rest B) New electrocardiographic changes suggestive of acute ischemia C) Typical rise and fall in cardiac biomarkers (refer to definition of spontaneous myocardial infarction).
  Probable stent thrombosis Regardless of the time after the index procedure, any myocardial infarction that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent/scaffold thrombosis and in the absence of any other obvious cause.
  Timing of ST (duration after stent implantation) Acute: 0-24 h & Sub-acute >24 h-30 d & Late >30 d-1 y & Very late >1 y

CONTACTS AND LOCATIONS:
Overall Officials: Magdy algowhary, MD, Principal Investigator — Assiut University Heart Hospital, Department of Cardiology, Assiut University, Assiut, Egypt.; Salwa R Demitry, MD, Principal Investigator — Assiut University Heart Hospital, Department of Cardiology, Assiut University, Assiut, Egypt.
Locations (1):
- Assiut, Asyut, Alsabeel, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valdes-Chavarri M, Kedev S, Neskovic AN, Moris de la Tassa C, Zivkovic M, Trillo Nouche R, Vazquez Gonzalez N, Bartorelli AL, Antoniucci D, Tamburino C, Colombo A, Abizaid AA, McFadden E, Garcia-Garcia HM, Milasinovic D, Stankovic G. Randomised evaluation of a novel biodegradable polymer-based sirolimus-eluting stent in ST-segment elevation myocardial infarction: the MASTER study. EuroIntervention. 2019 Apr 5;14(18):e1836-e1842. doi: 10.4244/EIJ-D-17-01087. PMID 29957593
- [Background] Bangalore S, Toklu B, Patel N, Feit F, Stone GW. Newer-Generation Ultrathin Strut Drug-Eluting Stents Versus Older Second-Generation Thicker Strut Drug-Eluting Stents for Coronary Artery Disease. Circulation. 2018 Nov 13;138(20):2216-2226. doi: 10.1161/CIRCULATIONAHA.118.034456. PMID 29945934
- [Background] Poder TG, Erraji J, Coulibaly LP, Koffi K. Percutaneous coronary intervention with second-generation drug-eluting stent versus bare-metal stent: Systematic review and cost-benefit analysis. PLoS One. 2017 May 12;12(5):e0177476. doi: 10.1371/journal.pone.0177476. eCollection 2017. PMID 28498849
- [Background] Abizaid A, Kedev S, Kedhi E, Talwar S, Erglis A, Hlinomaz O, Masotti M, Fath-Ordoubadi F, Lemos PA, Milewski K, Botelho R, Costa R, Bangalore S. Randomised comparison of a biodegradable polymer ultra-thin sirolimus-eluting stent versus a durable polymer everolimus-eluting stent in patients with de novo native coronary artery lesions: the meriT-V trial. EuroIntervention. 2018 Dec 7;14(11):e1207-e1214. doi: 10.4244/EIJ-D-18-00762. PMID 30222120